CLINICAL TRIAL: NCT05296785
Title: Management of Open Tibial Fractures With Bone Loss Using Monorail Fixator Over Intramedullary Nail
Brief Title: Evaluate Clinical and Radiological Outcomes After Limb Reconstruction Using Monorail Fixator Over Intramedullary Nailing in Tibial Open Fractures With Bone Loss
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Hossam Eldeen Ahmed Neyaz, principle investigator, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17200694
Record Dates: First submitted 2022-02-28; First posted 2022-03-25 (Actual); Last update posted 2022-04-06 (Actual); Status verified 2022-03

CONDITIONS: Open Fracture Tibia
MeSH Terms: interventions — Fracture Fixation, Intramedullary

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Participants (Other): patients undergoes intramedullary nail with Limb Reconstruction System
  Interventions: Procedure: intramedullary nail with Limb Reconstruction System

INTERVENTIONS:
Procedure: intramedullary nail with Limb Reconstruction System — bone transport by Limb Reconstruction System over intramedullary nail on fracture tibia

SUMMARY:
Road traffic accidents (RTA) is the most common cause of open fractures of long bones, increase in RTA leading to increase of complex non-unions incidence. the Participants are usually undergoing multiple surgeries for healing or to eradicate infection, which in turn leading to loss of bone and soft tissues and require skin grafting, muscle pedicle graft or bone grafting. Sometimes the Participants end up with deformity, limb length discrepancy, joints stiffness, disuse osteoporosis and muscle atrophy after management

ELIGIBILITY:
Inclusion Criteria:

* Age from 18-60 years old.
* Open Grade II, Open Grade III (a & b) diaphyseal fractures of Tibia (judged after primary and/or secondary to debridement).
* Bone defect < 10 cm.
* Patients with Injury severity score (ISS) < 17.

Exclusion Criteria:

* Massive bone defect > 10 cm.
* Patients with ISS > 17, polytrauma patient.
* Age < 18 years old or > 60 years old.
* Associated vascular injury ischemic limb.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-04-01 (Estimated); Primary Completion 2024-04-01 (Estimated); Study Completion 2025-02-01 (Estimated)

PRIMARY OUTCOMES:
ASAMI Scoring System | 1 year
  excellent : active , no limping good : active with one or more of : limp , stiffness , significant pain Fair : active with at least three of the following : limping , stiffness , significant pain , reflex sympathetic syndrome Poor : Inactive Failures : Amputations